CLINICAL TRIAL: NCT04594226
Title: Efficacy of Electroacupuncture Therapy in Patients With Postherpetic Neuralgia: a Multicentre Randomised Controlled Trial
Brief Title: Electroacupuncture Therapy for Treating Postherpetic Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Lishui Hospital of Traditional Chinese Medicine (Unknown); Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, Dexiong Han, Head of the Acupuncture Department, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019ZB057_
Record Dates: First submitted 2020-10-11; First posted 2020-10-20 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Postherpetic Neuralgia
Keywords: Electroacupuncture; Postherpetic neuralgia; Pain; Randomized controlled trial; Protocol
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA combined with medication group (Experimental): Patients in this group will receive electroacupuncture combined with gabapentin.
  Interventions: Procedure: EA combined with medication; Drug: Medication
- Medication group (Active Comparator): Participants in this group will only receive gabapentin.
  Interventions: Drug: Medication

INTERVENTIONS:
Procedure: EA combined with medication — Primary acupoints include Ashi points, Jiaji acupoints and Xi-cleft points. Jiaji points on the ipsilateral side will be selected according to the corresponding ganglia involved by HZ. Xi-cleft points will be selected based on the distribution regions of PHN. For pain sites that mainly distributed in the gallbladder meridian, GB36 will be selected. For pain sites that mainly distributed in the stomach meridian, ST34 will be selected. For pain sites that mainly distributed in the gallbladder meridian, BL63 will be selected. For pain sites that mainly distributed in the large intestine meridian, LI7 will be selected. Supplementary acupoints will be chosen based on TCM syndrome differentiation.
  Operation: Two paired of acupoints are connected to the EA apparatus. EA parameter is selected as 2/100Hz wave. EA intensity is selected according to the patients' endurance. Needles will be retained and EA will last for 30 mins for each session.
  Arms: EA combined with medication group
Drug: Medication — The dosage of gabapentin starts from 100mg Tid. 100mg-300mg can be increased every 3-7 days and taken in three doses, but the total amount is not more than 1800mg/day. The dosage of gabapentin will be adjusted according to the patient's condition until his pain is effectively controlled. After maintaining the medication for two weeks, the dosage can be gradually reduced and 100mg can be reduced every 3-7 days.

SUMMARY:
Postherpetic neuralgia (PHN) has a high incidence rate and severely impact on quality of life and health care costs, interfering with physical, emotional and social functioning of affected patients. Current therapeutic options for PHN mainly include analgetic and local anaesthesia for selective nerve blockade. Nevertheless, the efficacy of analgetic is always limited by inevitable side effects, in which patients have poor compliance. Moreover, for some most suffering patients, the control of pain is often unsatisfactory despite the administration of complex combinations. As a non-pharmarceutical therapy, acupuncture is widely use for a wide range of pain conditions. Thus, it might be an alternative treatment for PHN. The aim of this multicenter randomized controlled trial is to investigate the efficacy and safety of electroacupuncture therapy in patients with postherpetic neuralgia.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 132 patients with postherpetic neuralgia. All patients will be randomly assigned to either the EA combined with medication group or the medication group via a computerized central randomization system in a 1:1 ratio. Primary outcomes will be change in sensory thresholds and pain intensity. Secondary outcomes will be change in dosage of analgetic, quality of life, anxiety and depression severity and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have a medical history of herpes zoster;
2. Skin lesion has healed in the region of herpes zoster, but the duration of postherpetic neuralgia persist for more than 30 days.
3. 20 ≤ age ≤80 years, male or female
4. Participants can fully understand the study protocol and written informed consent is signed.

Exclusion Criteria:

1. Acute herpes zoster, herpes zoster has not disappeared;
2. Herpes zoster belongs to a special type, such as ophthalmic herpes zoster, auricular herpes zoster, HZ that involves internal organs, meningeal herpes zoster, and disseminated herpes zoster.
3. Pregnant or lactating women;
4. Patients have severe complications in cardiovascular, cerebrovascular, liver, kidney, hematopoietic and other systems,or have malignant tumor, mental illness, immune deficiency, hemorrhagic disorders and other diseases;
5. Patients have severe cognitive impairment and can not understand the study protocol;
6. Patients can not receive electroacupuncture treatment due to any reasons.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in sensory thresholds | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Sensory thresholds is measured by quantitative sensory testing
Change in pain intensity | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Pain intensity is measured by Zoster Brief Pain Inventory (ZBPI)

SECONDARY OUTCOMES:
Change in dosage of analgetic | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Dosage of analgetic
Change in score of quality of life | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Quality of life is measure by 36-item Short Form Health Survey (SF-36)
Change in score of anxiety and depression severity | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Anxiety and depression severity is measure by Hospital Anxiety and Depression Scale (HADS)
Change in score of sleep quality | before treatment, 2 weeks after treatment, 4 weeks after treatment, 6 weeks after treatment, at 8-week follow-up
  Sleep quality is measured by Pittsburgh Sleep Quality Index (PSQI)
Adverse events | Up to 6 weeks of treatment
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dexiong Han, M.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saguil A, Kane S, Mercado M, Lauters R. Herpes Zoster and Postherpetic Neuralgia: Prevention and Management. Am Fam Physician. 2017 Nov 15;96(10):656-663. PMID 29431387
- [Background] Johnson RW, Rice AS. Clinical practice. Postherpetic neuralgia. N Engl J Med. 2014 Oct 16;371(16):1526-33. doi: 10.1056/NEJMcp1403062. No abstract available. PMID 25317872
- [Background] Forbes HJ, Thomas SL, Smeeth L, Clayton T, Farmer R, Bhaskaran K, Langan SM. A systematic review and meta-analysis of risk factors for postherpetic neuralgia. Pain. 2016 Jan;157(1):30-54. doi: 10.1097/j.pain.0000000000000307. PMID 26218719
- [Background] Lin CS, Lin YC, Lao HC, Chen CC. Interventional Treatments for Postherpetic Neuralgia: A Systematic Review. Pain Physician. 2019 May;22(3):209-228. PMID 31151330
- [Background] Wang Y, Li W, Peng W, Zhou J, Liu Z. Acupuncture for postherpetic neuralgia: Systematic review and meta-analysis. Medicine (Baltimore). 2018 Aug;97(34):e11986. doi: 10.1097/MD.0000000000011986. PMID 30142834
- [Background] Avijgan M, Hajzargarbashi ST, Kamran A, Avijgan M. Postherpetic Neuralgia: Practical Experiences Return to Traditional Chinese Medicine. J Acupunct Meridian Stud. 2017 Jun;10(3):157-164. doi: 10.1016/j.jams.2017.02.003. Epub 2017 Feb 28. PMID 28712474
- [Background] Ruengwongroj P, Muengtaweepongsa S, Patumanond J, Phinyo P. Effectiveness of press needle treatment and electroacupuncture in patients with postherpetic neuralgia: A matched propensity score analysis. Complement Ther Clin Pract. 2020 Aug;40:101202. doi: 10.1016/j.ctcp.2020.101202. Epub 2020 May 25. PMID 32891279
- [Background] Zhang Y, Liang Z, Li S, Yang L, Guo T, Xu Y, Yang J, Xu Q, Zhang Q, Zhao J, Li C, Liu X. Fire needle plus cupping for acute herpes zoster: study protocol for a randomized controlled trial. Trials. 2020 Aug 6;21(1):701. doi: 10.1186/s13063-020-04599-2. PMID 32762718
- [Background] Wang L, Qiu L, Zheng X, Ouyang J, Zhang M, He L, Zeng S, Liu B, Peng J. Effectiveness of electroacupuncture at Jiaji acupoints (EX-B2), plus moxibustion and intermediate on postherpetic neuralgia: a randomized controlled trial. J Tradit Chin Med. 2020 Feb;40(1):121-127. PMID 32227773
- [Background] Pei W, Zeng J, Lu L, Lin G, Ruan J. Is acupuncture an effective postherpetic neuralgia treatment? A systematic review and meta-analysis. J Pain Res. 2019 Jul 16;12:2155-2165. doi: 10.2147/JPR.S199950. eCollection 2019. PMID 31410050
- [Background] Liu K, Zeng J, Pei W, Chen S, Luo Z, Lu L, Lin G. Assessing the reporting quality in randomized controlled trials of acupuncture for postherpetic neuralgia using the CONSORT statement and STRICTA guidelines. J Pain Res. 2019 Jul 29;12:2359-2370. doi: 10.2147/JPR.S210471. eCollection 2019. PMID 31534360
- [Derived] Hu H, Shen Y, Li X, Tian H, Li X, Li Y, Cheng Y, Wu L, Han D. Efficacy of Electroacupuncture Therapy in Patients With Postherpetic Neuralgia: Study Protocol for a Multicentre, Randomized, Controlled, Assessor-Blinded Trial. Front Med (Lausanne). 2021 May 21;8:624797. doi: 10.3389/fmed.2021.624797. eCollection 2021. PMID 34095161